CLINICAL TRIAL: NCT00335062
Title: TSH Receptor Antibody Heterogeneity in Children and Adolescents With Graves' Disease
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Rosalind Brown, Director of Clinical Trials, Boston Children's Hospital
Other Study IDs: S05-05-066
Record Dates: First submitted 2006-06-06; First posted 2006-06-08 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Graves' Disease
Keywords: Autoimmune thyroid disease; Children and Adolescents; TSH Receptor Antibodies
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Graves' disease, the most common form of hyperthyroidism in children, is caused by Thyrotropin (TSH) Receptor Antibodies (TRAbs) that mimic the action of TSH. The disease leads to significant morbidity in children both due to the prolonged course of antithyroid medication often required for sustained immunological remission and the high risk of relapse when medication is withdrawn. The ability to predict which patients are most likely to fail medical management would greatly improve the choice of therapy. In the past, large goiter size, age at diagnosis, increased biochemical severity, and decreased body mass index have all been associated with a poorer prognosis, but these clinical indicators lack sensitivity and specificity. Preliminary data suggest that the new TRAb assays are both sensitive and specific for the measurement of TRAbs in children with Graves' disease. In addition, variation in these antibodies over time is not the same in all patients. The goal of this proposal will be to prospectively follow children with newly diagnosed Graves' disease and use microarray technology to determine if there are genes whose expression differ in patients who respond to medical therapy versus those who will need more definitive therapy earlier in their disease.

DETAILED DESCRIPTION:
In the present grant proposal, we plan to utilize two new assays (binding and bioassay) in order to identify additional predictors of Graves' disease and apply them to a well characterized group of patients with Graves' disease followed prospectively. More specifically, we plan to further investigate the antibodies by measuring lambda: kappa light chain antibody ratios in pediatric patients. We will assess epitope heterogeneity by using novel chimeric proteins in which specific portions of the TSH receptor have been replaced with the closely related LH receptor. We will utilize microarray technology to determine if there are differences in gene expression profiles in responders versus non responders. It is hoped that these methods will lead to an improved ability to follow disease progression and to monitor efficacy of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-21 years
* Suppressed Thyroid Stimulating Hormone (TSH)
* Elevated Triiodothyronine (T3), Thyroxine (T4)

Exclusion Criteria:

* Pregnancy
* Toxic Nodule
* Currently receiving steroids or thyroid hormone replacement
* Bacterial, Viral, Radiation, or Autoimmune thyroiditis

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents referred to a tertiary medical center with hyperthyroidism.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2005-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the disappearance of TSH receptor Abs (as assessed by both ELISA and bioassay) from the circulation. | end of study

SECONDARY OUTCOMES:
2) The secondary outcome will be normalization of thyroid function tests (T4, free T4, Total T3, and TSH) on a low dose of Tapazole 2.5-5.0 mg per day. | end of study

OTHER OUTCOMES:
3) In the neonatal Graves' disease patient, the primary outcome will be the clearance of both TBII and TSI from the infant's sera (as assessed by both ELISA and bioassay). | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind S Brown, Principal Investigator — Children's Hosptial Boston/Harvard Medical School
Locations (1):
- Childrens' Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- See also: THYROID DISEASE MANAGER © offers an up-to-date analysis of thyrotoxicosis, hypothyroidism, thyroid nodules and cancer, thyroiditis, and all aspects of human thyroid disease. — http://www.thyroidmanager.org